CLINICAL TRIAL: NCT04537598
Title: Ultrasound Guided Continuous Erector Spinae Plane Block Versus Patient Controlled Analgesia in Patients Undergoing Nephrectomy for Renal Malignancies: A Randomized Controlled Study
Brief Title: Erector Spinae Plane Block for Post-nephrectomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ehab Hanafy Shaker, Assistant professor of Anesthesia, intensive care and pain releif, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESPB for nephrectomy
Record Dates: First submitted 2020-08-28; First posted 2020-09-03 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient controlled analgesia (Active Comparator): 30 patients will receive only postoperative IV PCA alone for postoperative analgesia.
  Interventions: Procedure: Morphine patient controlled analgesia
- Erector Spinae plane block (Active Comparator): 30 patients will receive continuous ESPB for postoperative analgesia.
  Interventions: Procedure: Erector Spinae plane block

INTERVENTIONS:
Procedure: Morphine patient controlled analgesia — 30 patients will receive PCA only for postoperative analgesia
  Arms: patient controlled analgesia
Procedure: Erector Spinae plane block — 30 patients will receive continuous ESPB for postoperative analgesia
  Arms: Erector Spinae plane block

SUMMARY:
Acute postoperative pain proper management is important not only for patient satisfaction but also for patient outcome. It may also predispose patients to chronic post-surgical pain .Open nephrectomy is still conducted, although the use of laparoscopic or robotic surgery has increased recently. A flank approach with an eleventh rib partial resection.Several modalities have been implemented for acute postoperative pain control. Intravenous (IV) opioids is one of the earliest and most widely used method, it is insufficient only for managing postoperative pain in some patients with severe pain besides their side effects.ESPB is a relatively simple technique with easily identified sonographic landmarks. Additionally, the ESPB has the potential to provide both somatic and visceral sensory blockade.The aim of this study is to evaluate the effect of ESPB in acute postoperative pain and opioid consumption in patients undergoing open nephrectomy in renal cancer patients.

DETAILED DESCRIPTION:
Acute postoperative pain proper management is important not only for patient satisfaction but also for patient outcome. In addition to its early effects, poorly controlled acute postoperative pain may predispose patients to chronic post-surgical pain.

Open nephrectomy is still conducted, although the use of laparoscopic or robotic surgery has increased recently. A flank approach with an eleventh rib partial resection, which is the main method for open nephrectomy at our institution, could make for better dissection of the renal pelvis and the pedicles, and provide the best circumstances for nephrectomy; however, it induces more persistent pain compared with other approaches.

Several modalities have been implemented for acute postoperative pain control. Intravenous (IV) opioids is one of the earliest and most widely used method, it is insufficient only for managing postoperative pain in some patients with severe pain. In addition, opioids have many side effects like respiratory depression, nausea, vomiting and constipation hence it is important to decrease opioids use and the transition to other modalities such as regional blocks, nerve blocks, NSAIDs and multimodalities.ESPB is a relatively simple technique with easily identified sonographic landmarks. Additionally, the ESPB has the potential to provide both somatic and visceral sensory blockade.

The erector spinae muscle (ESM) is a complex formed by the spinalis, longissimus thoracis, and iliocostalis muscles that run vertically in the back. The ESP block is performed by depositing the local anesthetic (LA) in the fascial plane, deeper than the ESM at the tip of the transverse process of the vertebra. Hence, LA is distributed in the cranio-caudal fascial plane.Additionally, it diffuses anteriorly to the paravertebral and epidural spaces, and laterally to the intercostal space at several levels.

There are different case studies about the use of erector spinae block in nephrectomy but there is no randomized controlled study about it until now so it will be one of the earliest studies that investigate the effect of ESPB to relief acute postoperative pain in patients undergoing open nephrectomy.

The aim of this study is to evaluate the effect of ESPB in acute postoperative pain and opioid consumption in patients undergoing open nephrectomy in renal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Physical status ASA II.
* Age ≥ 18 and ≤ 65 Years.
* Body mass index (BMI): > 20 kg/m2 and < 40 kg/m2.

Exclusion Criteria:

* Patient refusal
* Known sensitivity or contraindication to local anesthetics.
* History of psychological disorders.
* Localized infection at the site of block.

  * Coagulopathies with platelet count below 50,000 or an INR>1.5.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2022-05-28 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
measurement of visual analogue score | 1 week
  it is a scoring system from 0 to 100 mm where 100 represents the worst pain and 0 indicates no pain

CONTACTS AND LOCATIONS:
Overall Officials: Ehab H Gendy, MD, Principal Investigator — Assistant Professor of Anesthesia, intensive care and pain releif
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
we can share IPD after journal accepting the manuscript